CLINICAL TRIAL: NCT07228663
Title: Rivaroxaban Plus Acetylsalicylic Acid Versus Standard of Care for Arterial and Venous Cardiovascular Prevention After Hip Fracture Surgery in Patients With Myocardial Injury: a Pilot Randomized Trial
Brief Title: Hip Fracture Surgery Arterial and Venous Thrombotic Events Prevention
Acronym: HIPSTER-Pilot
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Venous Thromboembolism Clinical Trials and Outcomes Research (CanVECTOR) Network (Network); International Network of VENous Thromboembolism Clinical Research Networks (Unknown)
Responsible Party: Principal Investigator, Federico Germini, Associate Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HIPSTER-2024
Record Dates: First submitted 2025-08-16; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-08

CONDITIONS: Hip Fracture Surgery; Cardiovascular Prevention; Venous Thromboembolism (VTE)
Keywords: rivaroxaban; acetylsalicylic acid; cardiovascular prevention; hip fracture surgery; myocardial injury; venous thromboembolism (VTE)
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban; Aspirin; Dalteparin; Enoxaparin; Tinzaparin; Fondaparinux; N(4)-oleylcytosine arabinoside; apixaban

STUDY DESIGN:
Intervention Model Description: A total of 100 participants aged ≥45 years who received hip fracture surgery and experienced a myocardial injury will be randomized to receive either rivaroxaban 2.5 mg twice daily plus ASA 75-100 mg daily for 90 days or standard VTE prophylaxis with an anticoagulant for ~30 days, as per the standard of care.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Statisticians.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- rivaroxaban plus ASA (Active Comparator): rivaroxaban 2.5mg twice daily plus ASA 75-100mg daily for 90 days
  Interventions: Drug: rivaroxaban and ASA
- standard VTE prophylaxis with an anticoagulant (Active Comparator): Institution's standard of care for thromboprophylaxis with a low-dose anticoagulant for ~30 days (as per the standard of care). Regimens could include low-molecular-weight heparin, fondaparinux, or direct oral anticoagulant.
  Interventions: Drug: Low-molecular weight heparin; Drug: Fondaparinux; Drug: Direct Oral Anticoagulant (DOAC)

INTERVENTIONS:
Drug: rivaroxaban and ASA — rivaroxaban 2.5 mg orally BID and ASA 75-100 mg OD for 90 days
  Other Names: acetylsalicylic acid; Xarelto
  Arms: rivaroxaban plus ASA
Drug: Low-molecular weight heparin — Enoxaparin: 40 mg subcutaneously OD (or 30 mg subcutaneously BID); Dalteparin: 5000 IU subcutaneously OD (or alternative dosing based on institutional protocol); Tinzaparin: 4500 IU subcutaneous OD
  Other Names: enoxaparin; dalteparin; tinzaparin
  Arms: standard VTE prophylaxis with an anticoagulant
Drug: Fondaparinux — 2.5 mg subcutaneously OD
  Other Names: arixtra
  Arms: standard VTE prophylaxis with an anticoagulant
Drug: Direct Oral Anticoagulant (DOAC) — Rivaroxaban 10 mg OD or apixaban 2.5 mg BID, started after surgery or after a period of LMWH.
  Other Names: rivaroxaban; apixaban
  Arms: standard VTE prophylaxis with an anticoagulant

SUMMARY:
A third of patients undergoing surgery for a hip fracture develop a myocardial injury (i.e., an elevated troponin measurement), and these patients are at substantial risk of death and morbidity. Current prophylaxis strategies focus on preventing venous thromboembolism (VTE); however, arterial events are more common and carry a poor prognosis. The association of acetylsalicylic acid (ASA) 75-100 mg once daily and rivaroxaban 2.5 mg twice a day (the regimen used in the COMPASS trial) might prevent both VTE and arterial cardiovascular events. Among patients who have undergone hip fracture surgery and have evidence of myocardial injury, to explore the feasibility of a randomized controlled trial (RCT) comparing rivaroxaban 2.5 mg twice daily + low-dose ASA (75-100 mg) for 90 days, with standard VTE thromboprophylaxis for 30 days, for prevention of major cardiovascular events. The HIPSTER-Pilot is a multicenter, international, open-label, pilot RCT with blinded outcome adjudication. A total of 100 participants aged ≥45 years who received hip fracture surgery and experienced a myocardial injury will be randomized to receive either rivaroxaban 2.5 mg twice daily plus ASA 75-100 mg daily for 90 days or standard VTE prophylaxis with an anticoagulant for 30 days. The primary feasibility outcome will be the recruitment rate. Other feasibility measures include completeness of follow-up and adherence to the treatment. Exploratory clinical outcomes will be assessed. This pilot trial will provide information on the feasibility of conducting a larger RCT to evaluate the efficacy and safety of the COMPASS regimen for preventing arterial and venous thrombotic events after hip fracture surgery in patients who have had myocardial injury. The results of this feasibility study will inform the design of the full-scale trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥45 years, received surgery for a hip fracture due to a low-energy mechanism, and myocardial injury (i.e., an elevated troponin measurement).

Exclusion Criteria:

* Centers in which standard of care for VTE prophylaxis after hip fractures is ASA, alone or in combination with other drugs; patients with GFR <15mL/min; patients with drug interactions and conditions that prevent the use of the standard of care or intervention [Known allergy to the study drugs; pregnancy; an indication for anticoagulation, for dual antiplatelet therapy, for a P2Y12 inhibitor; already on rivaroxaban 2.5 mg twice daily + ASA before the fracture; bleeding diathesis that in the judgment of the investigator precludes the use of anticoagulant prophylaxis; history of significant hepatic disease (Child-Pugh B or C, see supplementary material) or any other condition that, in the judgment of the investigator, precludes the use of rivaroxaban; concomitant use of drugs that are strong inhibitors or strong inducers of P-glycoprotein (P-gp, e.g., systemic azole antimycotics, such as ketoconazole, and human immunodeficiency virus [HIV]-protease inhibitors, such as ritonavir) and/or Cytochrome P450 3A4 (CYP3A4)]; expected requirement for major surgery post-arthroplasty within 90 days; women Persons of childbearing potential who are not abstinent or do not use appropriate contraception or are breast-feeding; unable or unwilling to provide consent; previous participation in the HIPSTER trial; participation in another anticoagulant or antiplatelet study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Through study completion, an average of 1 year.
  Number of patients recruited per month per site

SECONDARY OUTCOMES:
FUP completion | assessed at 30 and 90 days
  Proportion of patients with a complete follow up
Treatment adherence | 30 and 90 days for the intervention, pre-specified treatment duration as per standard of care for the control.
  Proportion of number of days on treatment

OTHER OUTCOMES:
all-cause mortality, MI, non-hemorrhagic stroke, peripheral arterial thrombosis, and symptomatic objectively confirmted VTE | From randomization to 90 days post-randomization.
  Composite. Also each individual component will be assessed.
Cardiovascular mortality | From randomization to 90 days post-randomization.
Major bleeding events | From randomization to 90 days post-randomization.
  Major bleeding events as defined by the ISTH.
Clinically relevant nonmajor bleeding | From randomization to 90 days post-randomization.
Minor bleeding | From randomization to 90 days post-randomization.
Bleeding independently associated with mortality after non-cardiac surgery (BIMS) | From randomization to 90 days post-randomization.
  Bleeding leading to a postoperative haemoglobin <70 g/L, transfusion of 1 unit of red blood cells, or bleeding that was judged to be the cause of death.
Quality of life (EQ-5D-5L) | 90 days
  Measured with EQ-5D-5L
Hospitalizations | From randomization to 90-days post randomization.
  The length of stay and re-hospitalizations as measures of resource utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Germini, Doctor of Medicine, Principal Investigator — McMaster University
Locations (3):
- Canada (2):
  - St.Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario
- Humanitas Research Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Available to share upon reasonable request, but will likely not unblind before completing a full-scale trial.

REFERENCES:
- [Background] Anderson DR, Dunbar M, Murnaghan J, Kahn SR, Gross P, Forsythe M, Pelet S, Fisher W, Belzile E, Dolan S, Crowther M, Bohm E, MacDonald SJ, Gofton W, Kim P, Zukor D, Pleasance S, Andreou P, Doucette S, Theriault C, Abianui A, Carrier M, Kovacs MJ, Rodger MA, Coyle D, Wells PS, Vendittoli PA. Aspirin or Rivaroxaban for VTE Prophylaxis after Hip or Knee Arthroplasty. N Engl J Med. 2018 Feb 22;378(8):699-707. doi: 10.1056/NEJMoa1712746. PMID 29466159
- [Background] Schulman S, Angeras U, Bergqvist D, Eriksson B, Lassen MR, Fisher W; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in surgical patients. J Thromb Haemost. 2010 Jan;8(1):202-4. doi: 10.1111/j.1538-7836.2009.03678.x. Epub 2009 Oct 30. PMID 19878532
- [Background] Roshanov PS, Eikelboom JW, Sessler DI, Kearon C, Guyatt GH, Crowther M, Tandon V, Borges FK, Lamy A, Whitlock R, Biccard BM, Szczeklik W, Panju M, Spence J, Garg AX, McGillion M, VanHelder T, Kavsak PA, de Beer J, Winemaker M, Le Manach Y, Sheth T, Pinthus JH, Siegal D, Thabane L, Simunovic MRI, Mizera R, Ribas S, Devereaux PJ. Bleeding Independently associated with Mortality after noncardiac Surgery (BIMS): an international prospective cohort study establishing diagnostic criteria and prognostic importance. Br J Anaesth. 2021 Jan;126(1):163-171. doi: 10.1016/j.bja.2020.06.051. Epub 2020 Aug 5. PMID 32768179
- [Background] Avery KN, Williamson PR, Gamble C, O'Connell Francischetto E, Metcalfe C, Davidson P, Williams H, Blazeby JM; members of the Internal Pilot Trials Workshop supported by the Hubs for Trials Methodology Research. Informing efficient randomised controlled trials: exploration of challenges in developing progression criteria for internal pilot studies. BMJ Open. 2017 Feb 17;7(2):e013537. doi: 10.1136/bmjopen-2016-013537. PMID 28213598
- [Background] National Guideline Centre (UK). Venous thromboembolism in over 16s: Reducing the risk of hospital-acquired deep vein thrombosis or pulmonary embolism. London: National Institute for Health and Care Excellence (NICE); 2018 Mar. Available from http://www.ncbi.nlm.nih.gov/books/NBK493720/ PMID 29697228
- [Background] Halvorsen S, Mehilli J, Cassese S, Hall TS, Abdelhamid M, Barbato E, De Hert S, de Laval I, Geisler T, Hinterbuchner L, Ibanez B, Lenarczyk R, Mansmann UR, McGreavy P, Mueller C, Muneretto C, Niessner A, Potpara TS, Ristic A, Sade LE, Schirmer H, Schupke S, Sillesen H, Skulstad H, Torracca L, Tutarel O, Van Der Meer P, Wojakowski W, Zacharowski K; ESC Scientific Document Group. 2022 ESC Guidelines on cardiovascular assessment and management of patients undergoing non-cardiac surgery. Eur Heart J. 2022 Oct 14;43(39):3826-3924. doi: 10.1093/eurheartj/ehac270. No abstract available. PMID 36017553
- [Background] Duceppe E, Parlow J, MacDonald P, Lyons K, McMullen M, Srinathan S, Graham M, Tandon V, Styles K, Bessissow A, Sessler DI, Bryson G, Devereaux PJ. Canadian Cardiovascular Society Guidelines on Perioperative Cardiac Risk Assessment and Management for Patients Who Undergo Noncardiac Surgery. Can J Cardiol. 2017 Jan;33(1):17-32. doi: 10.1016/j.cjca.2016.09.008. Epub 2016 Oct 4. PMID 27865641
- [Background] Devereaux PJ, Marcucci M, Painter TW, Conen D, Lomivorotov V, Sessler DI, Chan MTV, Borges FK, Martinez-Zapata MJ, Wang CY, Xavier D, Ofori SN, Wang MK, Efremov S, Landoni G, Kleinlugtenbelt YV, Szczeklik W, Schmartz D, Garg AX, Short TG, Wittmann M, Meyhoff CS, Amir M, Torres D, Patel A, Duceppe E, Ruetzler K, Parlow JL, Tandon V, Fleischmann E, Polanczyk CA, Lamy A, Astrakov SV, Rao M, Wu WKK, Bhatt K, de Nadal M, Likhvantsev VV, Paniagua P, Aguado HJ, Whitlock RP, McGillion MH, Prystajecky M, Vincent J, Eikelboom J, Copland I, Balasubramanian K, Turan A, Bangdiwala SI, Stillo D, Gross PL, Cafaro T, Alfonsi P, Roshanov PS, Belley-Cote EP, Spence J, Richards T, VanHelder T, McIntyre W, Guyatt G, Yusuf S, Leslie K; POISE-3 Investigators. Tranexamic Acid in Patients Undergoing Noncardiac Surgery. N Engl J Med. 2022 May 26;386(21):1986-1997. doi: 10.1056/NEJMoa2201171. Epub 2022 Apr 2. PMID 35363452
- [Background] Douketis JD, Spyropoulos AC, Murad MH, Arcelus JI, Dager WE, Dunn AS, Fargo RA, Levy JH, Samama CM, Shah SH, Sherwood MW, Tafur AJ, Tang LV, Moores LK. Perioperative Management of Antithrombotic Therapy: An American College of Chest Physicians Clinical Practice Guideline. Chest. 2022 Nov;162(5):e207-e243. doi: 10.1016/j.chest.2022.07.025. Epub 2022 Aug 11. PMID 35964704
- [Background] Sheth T, Natarajan MK, Hsieh V, Valettas N, Rokoss M, Mehta S, Jolly S, Tandon V, Bezerra H, Devereaux PJ. Incidence of thrombosis in perioperative and non-operative myocardial infarction. Br J Anaesth. 2018 Apr;120(4):725-733. doi: 10.1016/j.bja.2017.11.063. Epub 2017 Nov 21. PMID 29576113
- [Background] Bonaca MP, Bauersachs RM, Anand SS, Debus ES, Nehler MR, Patel MR, Fanelli F, Capell WH, Diao L, Jaeger N, Hess CN, Pap AF, Kittelson JM, Gudz I, Matyas L, Krievins DK, Diaz R, Brodmann M, Muehlhofer E, Haskell LP, Berkowitz SD, Hiatt WR. Rivaroxaban in Peripheral Artery Disease after Revascularization. N Engl J Med. 2020 May 21;382(21):1994-2004. doi: 10.1056/NEJMoa2000052. Epub 2020 Mar 28. PMID 32222135
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Background] Eikelboom JW, Connolly SJ, Bosch J, Dagenais GR, Hart RG, Shestakovska O, Diaz R, Alings M, Lonn EM, Anand SS, Widimsky P, Hori M, Avezum A, Piegas LS, Branch KRH, Probstfield J, Bhatt DL, Zhu J, Liang Y, Maggioni AP, Lopez-Jaramillo P, O'Donnell M, Kakkar AK, Fox KAA, Parkhomenko AN, Ertl G, Stork S, Keltai M, Ryden L, Pogosova N, Dans AL, Lanas F, Commerford PJ, Torp-Pedersen C, Guzik TJ, Verhamme PB, Vinereanu D, Kim JH, Tonkin AM, Lewis BS, Felix C, Yusoff K, Steg PG, Metsarinne KP, Cook Bruns N, Misselwitz F, Chen E, Leong D, Yusuf S; COMPASS Investigators. Rivaroxaban with or without Aspirin in Stable Cardiovascular Disease. N Engl J Med. 2017 Oct 5;377(14):1319-1330. doi: 10.1056/NEJMoa1709118. Epub 2017 Aug 27. PMID 28844192
- [Background] Devereaux PJ, Mrkobrada M, Sessler DI, Leslie K, Alonso-Coello P, Kurz A, Villar JC, Sigamani A, Biccard BM, Meyhoff CS, Parlow JL, Guyatt G, Robinson A, Garg AX, Rodseth RN, Botto F, Lurati Buse G, Xavier D, Chan MT, Tiboni M, Cook D, Kumar PA, Forget P, Malaga G, Fleischmann E, Amir M, Eikelboom J, Mizera R, Torres D, Wang CY, VanHelder T, Paniagua P, Berwanger O, Srinathan S, Graham M, Pasin L, Le Manach Y, Gao P, Pogue J, Whitlock R, Lamy A, Kearon C, Baigent C, Chow C, Pettit S, Chrolavicius S, Yusuf S; POISE-2 Investigators. Aspirin in patients undergoing noncardiac surgery. N Engl J Med. 2014 Apr 17;370(16):1494-503. doi: 10.1056/NEJMoa1401105. Epub 2014 Mar 31. PMID 24679062
- [Background] Devereaux PJ, Duceppe E, Guyatt G, Tandon V, Rodseth R, Biccard BM, Xavier D, Szczeklik W, Meyhoff CS, Vincent J, Franzosi MG, Srinathan SK, Erb J, Magloire P, Neary J, Rao M, Rahate PV, Chaudhry NK, Mayosi B, de Nadal M, Iglesias PP, Berwanger O, Villar JC, Botto F, Eikelboom JW, Sessler DI, Kearon C, Pettit S, Sharma M, Connolly SJ, Bangdiwala SI, Rao-Melacini P, Hoeft A, Yusuf S; MANAGE Investigators. Dabigatran in patients with myocardial injury after non-cardiac surgery (MANAGE): an international, randomised, placebo-controlled trial. Lancet. 2018 Jun 9;391(10137):2325-2334. doi: 10.1016/S0140-6736(18)30832-8. PMID 29900874
- [Background] Prevention of pulmonary embolism and deep vein thrombosis with low dose aspirin: Pulmonary Embolism Prevention (PEP) trial. Lancet. 2000 Apr 15;355(9212):1295-302. PMID 10776741
- [Background] Anderson DR, Morgano GP, Bennett C, Dentali F, Francis CW, Garcia DA, Kahn SR, Rahman M, Rajasekhar A, Rogers FB, Smythe MA, Tikkinen KAO, Yates AJ, Baldeh T, Balduzzi S, Brozek JL, Ikobaltzeta IE, Johal H, Neumann I, Wiercioch W, Yepes-Nunez JJ, Schunemann HJ, Dahm P. American Society of Hematology 2019 guidelines for management of venous thromboembolism: prevention of venous thromboembolism in surgical hospitalized patients. Blood Adv. 2019 Dec 10;3(23):3898-3944. doi: 10.1182/bloodadvances.2019000975. PMID 31794602
- [Background] Gao Y, Long A, Xie Z, Meng Y, Tan J, Lv H, Zhang L, Zhang L, Tang P. The compliance of thromboprophylaxis affects the risk of venous thromboembolism in patients undergoing hip fracture surgery. Springerplus. 2016 Aug 18;5(1):1362. doi: 10.1186/s40064-016-2724-1. eCollection 2016. PMID 27588255
- [Background] HIP ATTACK Investigators. Accelerated surgery versus standard care in hip fracture (HIP ATTACK): an international, randomised, controlled trial. Lancet. 2020 Feb 29;395(10225):698-708. doi: 10.1016/S0140-6736(20)30058-1. Epub 2020 Feb 9. PMID 32050090
- [Background] Gundel O, Thygesen LC, Gogenur I, Ekeloef S. Postoperative mortality after a hip fracture over a 15-year period in Denmark: a national register study. Acta Orthop. 2020 Feb;91(1):58-62. doi: 10.1080/17453674.2019.1680485. Epub 2019 Oct 22. PMID 31635502
- [Background] Sullivan KJ, Husak LE, Altebarmakian M, Brox WT. Demographic factors in hip fracture incidence and mortality rates in California, 2000-2011. J Orthop Surg Res. 2016 Jan 8;11:4. doi: 10.1186/s13018-015-0332-3. PMID 26746904
- [Background] Leslie WD, O'Donnell S, Lagace C, Walsh P, Bancej C, Jean S, Siminoski K, Kaiser S, Kendler DL, Jaglal S; Osteoporosis Surveillance Expert Working Group. Population-based Canadian hip fracture rates with international comparisons. Osteoporos Int. 2010 Aug;21(8):1317-22. doi: 10.1007/s00198-009-1080-1. Epub 2009 Oct 3. PMID 19802507
- [Background] Johnell O, Kanis JA. An estimate of the worldwide prevalence and disability associated with osteoporotic fractures. Osteoporos Int. 2006 Dec;17(12):1726-33. doi: 10.1007/s00198-006-0172-4. Epub 2006 Sep 16. PMID 16983459
- See also: Regulatory Decision Summary for Xarelto - Drug and Health Products Portal — https://dhpp.hpfb-dgpsa.ca/review-documents/resource/RDS00781
- See also: Xarelto | European Medicines Agency (EMA) — https://www.ema.europa.eu/en/medicines/human/EPAR/xarelto#authorisation-details
- See also: Food and Drug Administration (FDA). XARELTO (rivaroxaban) Label — https://www.accessdata.fda.gov/drugsatfda_docs/label/2021/215859s000lbl.pdf

DOCUMENTS (2):
  • Study Protocol (2025-06-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT07228663/Prot_000.pdf
  • Informed Consent Form (2025-06-09): https://cdn.clinicaltrials.gov/large-docs/63/NCT07228663/ICF_001.pdf